CLINICAL TRIAL: NCT02756390
Title: CBTI-CS: A Novel Cognitive-Behavioral Treatment for Insomnia in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Recklitis, Ph.D, Christopher Recklitis, PhD, MPH, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-336; R03CA201459-01 (NIH)
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Insomnia
Keywords: Insomnia cancer Survivor
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Sleep Hygiene & CBTI-CS) (Experimental): Participants receive a single educational session describing principles of Sleep Hygiene for Cancer Survivors. Those who continue to have significant symptoms of insomnia then receive 3 groups CBTI-CS sessions
  Interventions: Behavioral: CBTI-CS; Behavioral: Sleep Hygiene
- Arm B (Telehealth Pilot of CBTI-CS) (Other): Descriptive data collected on 10 participants (non-randomized) receiving CBTI-CS via Telehealth.
  Interventions: Behavioral: CBTI-CS via Telehealth

INTERVENTIONS:
Behavioral: CBTI-CS — CBTI-CS is a multi-modal intervention designed to address both cognitive and behavioral factors that perpetuate insomnia. Cognitive factors are addressed via cognitive restructuring and psychoeducation. Behavioral factors are addressed by structured sleep restriction, stimulus control and sleep hygiene techniques. Cancer treatment late-effects affecting sleep are addressed as potential contributors to these cognitive and behavioral factors, and as symptoms that may benefit from referral for medical evaluation/management. Participants are instructed in these cognitive-behavioral strategies as a group, but using analysis of personal sleep-log data, symptom self-reports and targeted workbook exercises, they are helped to tailor the intervention to address their specific needs.
  Other Names: Cognitive Behavioral Therapy for Insomnia -Cancer Survivors
  Arms: Arm A (Sleep Hygiene & CBTI-CS)
Behavioral: Sleep Hygiene — Education on health behaviors, sleep habits and environmental practices intended to promote good quality sleep. Recommendations target exercise and natural light exposure,use of stimulants and alcohol, daytime napping, timing of meals, creating a comfortable non-stimulating sleep space, and creating sleep rituals.
  Arms: Arm A (Sleep Hygiene & CBTI-CS)
Behavioral: CBTI-CS via Telehealth — The CBTI-CS intervention, a multi-modal intervention designed to address both cognitive and behavioral factors that perpetuate insomnia, will be administered via live video. conferencing. Participants will have a single in-person training session and subsequent CBTI-CS group sessions will be conducted by live video conference.
  Arms: Arm B (Telehealth Pilot of CBTI-CS)

SUMMARY:
This research study is evaluating the effectiveness of a 3-session behavioral intervention for insomnia in cancer survivors. This is a behavioral intervention study, and no medications are involved.

DETAILED DESCRIPTION:
This study is being done to test the usefulness of a 3-session cognitive-behavioral intervention for improving insomnia in cancer survivors. In this study, the investigators are testing whether this 3-session intervention (Cognitive Behavior Therapy for Insomnia in Cancer Survivors: CBTI-CS) will improve insomnia in cancer survivors whose continue to have insomnia symptoms after receiving sleep hygiene education.

In addition to the participants who will be offered sleep hygiene education and the 3-session CBTI-CS,10 additional participants will be recruited to participate in a pilot evaluation of the CBTI-CS intervention delivered via telehealth. This will be a pilot aspect of the study and data from these participants will be for descriptive purposes.

ELIGIBILITY:
Inclusion Criteria:

-≥ 18 years of age

* History of a cancer diagnosis
* No active cancer therapy (excluding chemoprevention) in the past year, and no cancer therapy planned in the next 6 months
* No surgery planned in the next 6 months
* Significant insomnia as evidenced by an Insomnia Severity Index score ≥12
* Able to read and write in English
* Willing to attend study group sessions
* Motivated and able to follow the demands of the CBTI-CS program, to keep sleep records, complete self-report symptom reports and make changes in their sleep schedule, including restricting their sleep.

Exclusion Criteria:

* Survivors who report ever being diagnosed with Bipolar Disorder will be excluded.
* Survivors who report ever being diagnosed with a Seizure Disorder or have experienced a seizure in the past 12 months will be excluded.
* Intention to adjust (decrease or increase) use of sedative, hypnotic, or over-the-counter medications that can affect sleep during the study period.
* Have diagnosed, untreated sleep apnea, or sleep apnea suspected by a physician but which has not been evaluated, or other sleep disorder
* Employment that involves irregular sleep patterns, such as shift-work or frequent long-distance travel that involves adjusting to different time zones, or employment in a position that could impact public safety (such as operating heavy machinery)
* Refusal to modify or reduce excessive alcohol use that is likely to interfere with an individual's sleep.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-12; Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
The Insomnia Severity Index (ISI) | Change from Baseline to 4-weeks post-intervention
  The ISI is a 7-item self-report questionnaire assessing severity, and impact of insomnia symptoms.

SECONDARY OUTCOMES:
Profile of Mood States - Short Form (POMS-SF) | Change from Baseline to 4 & 8 weeks post-intervention
  A 35-item measure which assesses mood states along several dimensions including Total Mood Disturbance.
The Insomnia Severity Index (ISI) | Change from Baseline to 8 weeks post-intervention
  The ISI is a 7-item self-report questionnaire assessing severity, and impact of insomnia symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Recklitis, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou ES, Partridge AH, Recklitis CJ. A pilot trial of brief group cognitive-behavioral treatment for insomnia in an adult cancer survivorship program. Psychooncology. 2017 Jun;26(6):843-848. doi: 10.1002/pon.4096. Epub 2016 Feb 12. PMID 26872123